Ethical Approval Code: 2016\_12\_09\_EHS



## Statistical Plan

## The Effect of Milk-Derived Protein Supplementation on the Recovery of Muscle Function following Resistance Exercise

## **Research Question or hypothesis:**

Ho: The type of protein beverage consumed following resistance exercise training will not affect the temporal

recovery of muscle function.



**Brief Background:** Resistance exercise can induce low-level muscle damage in conjunction with impaired contractile function. Milk-derived proteins contain, or induce, bioactive properties for muscle recovery.

Study Design: A block randomised, crossover design of 3 groups of 8 subjects per group

Participants: 24 young, healthy, resistance exercise trained, males aged 18 - 35 years.

**Statistical Analysis:** 

Independent variables: Dependent variables

TIME [9] MUSCLE FUNCTION [3]

Day 9,10,11,12,1,31,4,15,16,17 Maximal voluntary contraction (MVC)
Time to peak tension (TPT)

PROTEIN [3] 1-REP max lift (1RM)

MODEL: Mixed model analysis of variance

WPC-80, UL\_209, IsoN

- a. Within-subject factor, TIME (9)
- b. Between-subject factor, PROTEIN (3)
- c. Bonferroni corrected post-hoc comparisons

Ethical Approval Code: 2016\_12\_09\_EHS

- i. Graded effect sizes for mixed-model  $(\omega_p^2)$ , between-within subject, effects  $(\omega^2, d)$  reported alongside P-values  $(\alpha = 0.05)$
- ii. Violation to normality (Shapiro Wilk) data will be transformed by rank for analysis
- iii. Violation to homogeneity of variance-covariance matrices (Mauchly's W), e correction factors (Green-House Geisser, Huynh-Feld) will be applied
- iv. Violation to homogeneity of variance for post-hoc analysis (Levene's or Brown-Forsythe Test), Welsch-Satterthwaite corrections will be applied.